CLINICAL TRIAL: NCT02813694
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy Study to Compare the Efficacy and Safety of Oral Lefamulin (BC 3781) Versus Oral Moxifloxacin in Adults With Community-Acquired Bacterial Pneumonia
Brief Title: Study to Compare Lefamulin to Moxifloxacin for the Treatment of Adults With Pneumonia
Acronym: LEAP2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAB-BC-3781-3102
Record Dates: First submitted 2016-06-20; First posted 2016-06-27 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Community Acquired Pneumonia
Keywords: Pneumonia; CABP; CAP; Community acquired bacterial pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — lefamulin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lefamulin (Experimental): oral lefamulin, 600mg
  Interventions: Drug: lefamulin
- Moxifloxacin (Active Comparator): oral moxifloxacin, 400mg
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: lefamulin — antibacterial agent
  Other Names: BC-3781
  Arms: lefamulin
Drug: Moxifloxacin — antibacterial agent
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
This study evaluates the safety and efficacy of lefamulin, a pleuromutilin, for the treatment of adults with moderate community-acquired bacterial pneumonia

DETAILED DESCRIPTION:
Lefamulin is a potent, semi-synthetic antibacterial belonging to a novel class known as the pleuromutilins. The oral dosage form of lefamulin is under investigation in this study. Lefamulin's in vitro antibacterial profile includes the most important bacterial pathogens causing respiratory tract infection (RTI). The antibacterial spectrum comprises S. pneumoniae, H. influenzae, M. catarrhalis, the atypical respiratory pathogens L. pneumophila, C. pneumoniae, and M. pneumoniae, S. aureus including MRSA and CA-MRSA, ß-haemolytic streptococci including S. pyogenes and S. agalactiae, and Enterococcus faecium including vancomycin-resistant enterococci (VRE). Moreover, as demonstrated in cross-resistance studies, lefamulin remains active against clinical isolates resistant to the following antimicrobial(s) (classes): macrolides, lincosamides, streptogramin B, oxazolidinones, tetracyclines, ß lactams, quinolones, trimethoprim-sulfametoxazole, mupirocin, and vancomycin.

ELIGIBILITY:
Inclusion Criteria:

Each subject must:

1. Be male or female at least 18 years of age.
2. Provide written informed consent and be willing and able to adhere to the study-specified procedures and restrictions.
3. Have an acute illness (less than or equal to 7 days duration) with at least 3 of the following symptoms consistent with a lower respiratory tract infection (new or worsening):

   * Dyspnea.
   * New or increased cough.
   * Purulent sputum production.
   * Chest pain due to pneumonia.
4. Have at least 2 of the following vital sign abnormalities:

   * Fever (body temperature > 38.0 °C (100.4 °F) measured orally or equivalent temperature from an alternate body site) or hypothermia (body temperature < 35.0 °C (95.0 °F) measured orally or equivalent temperature from an alternate body site).
   * Hypotension (systolic blood pressure < 90 mmHg).
   * Tachycardia (heart rate > 100 beats/min).
   * Tachypnea (respiratory rate > 20 breaths/min).
5. Have at least 1 other clinical sign or laboratory finding of CABP:

   * Hypoxemia (i.e., O2 saturation < 90 % on room air or while receiving supplemental oxygen at subject's baseline requirement or PaO2 < 60 mmHg).
   * Auscultatory and/or percussion findings consistent with pneumonia (e.g., crackles, egophony, dullness).
   * White blood cell (WBC) count > 10 000 cells/mm3 or < 4 500 cells/mm3 or >15 % immature neutrophils (bands) regardless of total WBC count.
6. Have radiographically-documented pneumonia within 48 hours before enrollment (i.e., infiltrates in a lobar or multilobar distribution or diffuse opacities on chest x-ray or chest computed tomography scan consistent with acute bacterial pneumonia).
7. Have a Pneumonia Outcomes Research Team (PORT) Risk Class of II, III, or IV and be an appropriate candidate for oral antibiotic therapy as treatment for the current episode of CABP.

Exclusion Criteria:

Each subject must NOT:

1. Have received more than a single dose of a short-acting oral or IV antibacterial for CABP within 72 hours before randomization.
2. Require concomitant systemic antibacterial therapy potentially effective against CABP pathogens.
3. Have been hospitalized for 2 or more days within 90 days prior to the onset of symptoms or have resided in a nursing home or long-term healthcare facility within 30 days prior to the onset of symptoms. NOTE: Residence in an independent living facility is permitted.
4. Have confirmed or suspected CABP caused by a pathogen known to be resistant to any of the study drugs (e.g., MRSA, Pseudomonas aeruginosa, any pathogen of the Enterobacteriaceae Family) or attributable to etiologies other than community acquired bacterial pathogens (e.g., ventilator associated pneumonia, hospital acquired bacterial pneumonia, bacterial aspiration pneumonia, Pneumocystis jiroveci pneumonia or other fungal pneumonia, viral or mycobacterial infection of the lung).
5. Have a noninfectious cause of pulmonary infiltrates (e.g., pulmonary embolism, chemical pneumonitis from aspiration, hypersensitivity pneumonia, congestive heart failure, bronchial obstruction, lung cancer, cystic fibrosis).
6. Have confirmed or suspected pleural empyema (does not include sterile parapneumonic effusions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Gasink, MD, Study Chair — Nabriva Therapeutics AG
Locations (155):
- United States (25):
  - 1080, Beverly Hills, California
  - Site 1065, Fresno, California
  - 1078, Northridge, California
  - Site 1072, Oxnard, California
  - Site 1070, Sacramento, California
  - 1079, Sherman Oaks, California
  - Site 1053, Sylmar, California
  - Site 1064, DeBary, Florida
  - Site 1052, DeLand, Florida
  - 1076, Miami, Florida
  - Site 1051, Michigan City, Indiana
  - Site 1057, Natchitoches, Louisiana
  - Site 1073, New Bedford, Massachusetts
  - Site 1055, Detroit, Michigan
  - Site 1062, Detroit, Michigan
  - Site 1068, Royal Oak, Michigan
  - Site 1058, St Louis, Missouri
  - Site 1054, Butte, Montana
  - Site 1067, Lima, Ohio
  - Site 1056, Rapid City, South Dakota
  - 1077, Hendersonville, Tennessee
  - Site 1060, Houston, Texas
  - Site 1069, Houston, Texas
  - Site 1066, Splendora, Texas
  - Site 1059, Charlottesville, Virginia
- Argentina (8):
  - Site 3056, Buenos Aires
  - Site 3059, Buenos Aires AV
  - Site 3054, Córdoba
  - Site 3052, Córdoba
  - Site 3057, Córdoba
  - Site 3058, General Pacheco
  - Site 3051, La Plata
  - Site 3053, La Plata
- Brazil (3):
  - Site 3154, Belo Horizonte
  - Site 3153, Passo Fundo
  - Site 3152, São José do Rio Preto
- Bulgaria (13):
  - 4162, Rousse
  - Site 4154, Sliven
  - Site 4160, Sofia
  - Site 4157, Sofia
  - Site 4153, Sofia
  - Site 4156, Sofia
  - Site 4161, Sofia
  - 4163, Sofia
  - 4164, Sofia
  - 4165, Sofia
  - Site 4158, Stara Zagora
  - Site 4159, Vidin
  - Site 4152, Vratsa
- Chile (6):
  - Site 3353, Santiago
  - Site 3356, Santiago
  - Site 3357, Santiago
  - Site 3354, Talca
  - Site 3352, Temuco
  - Site 3355, Valdivia
- Georgia (5):
  - Site 4256, Batumi
  - Site 4253, Tbilisi
  - Site 4255, Tbilisi
  - Site 4252, Tbilisi
  - Site 4254, Tbilisi
- Hungary (4):
  - Site 4354, Budapest
  - Site 4353, Budapest
  - Site 4352, Mátraháza
  - Site 4351, Törökbálint
- Latvia (3):
  - Site 4451, Liepāja
  - Site 4453, Riga
  - Site 4452, Valmiera
- Mexico (4):
  - Site 1153, Aguascalientes
  - Site 1154, Guadalajara
  - Site 1151, Monterrey
  - Site 1152, Toluca
- Peru (15):
  - Site 3264, Grau, Lima region
  - Site 3262, Arequipa
  - Site 3263, Cusco
  - Site 3261, Cuzco
  - Site 3254, Ica
  - Site 3259, Iquitos
  - Site 3251, La Libertad
  - Site 3252, Lima
  - Site 3253, Lima
  - Site 3255, Lima
  - Site 3257, Lima
  - Site 3260, Lima
  - Site 3265, Lima
  - Site 3258, Lima Lima
  - Site 3256, Piura
- Philippines (6):
  - Site 2053, Caloocan
  - Site 2055, Cebu
  - Site 2052, Iloilo City
  - Site 2054, Quezon
  - Site 2056, Quezon City
  - Site 2051, Quezon City
- Poland (5):
  - Site 4755, Bochnia
  - Site 4754, Chodzież
  - Site 4753, Krakow
  - Site 4756, Krakow
  - Site 4757, Siedlce
- Romania (7):
  - Site 4855, Bucharest
  - Site 4858, Bucharest
  - Site 4854, Bucharest
  - Site 4853, Cluj-Napoca
  - Site 4851, Codlea
  - Site 4857, Craiova
  - Site 4856, Timișoara
- Russia (8):
  - Site 4953, Barnaul
  - Site 4957, Moscow
  - Site 4952, Moscow
  - Site 4954, Novosibirsk
  - Site 4955, Saint Petersburg
  - Site 4951, Saint Petersburg
  - Site 4959, Saratov
  - Site 4958, Smolensk
- Serbia (7):
  - Site 5052, Belgrade
  - Site 5056, Belgrade
  - Site 5051, Belgrade
  - 5057, Belgrade
  - Site 5053, Kamenitz
  - Site 5055, Knez-Selo
  - Site 5054, Kragujevac
- South Africa (6):
  - Site 5151, Bloemfontein
  - Site 5154, Krugersdorp
  - Site 5155, Middelburg
  - Site 5156, Pretoria
  - Site 5152, Queenswood
  - Site 5153, Witbank
- South Korea (7):
  - Site 2254, Uijeongbu-si, Gyeonggi-do
  - Site 2257, Bucheon-si
  - Site 2253, Daegu
  - Site 2255, Seoul
  - Site 2256, Seoul
  - Site 2251, Seoul
  - Site 2252, Seoul
- Spain (6):
  - Site 4554, Alicante
  - Site 4556, Badalona
  - Site 4552, Barcelona
  - Site 4555, Barcelona
  - Site 4553, Madrid
  - Site 4551, Madrid
- Taiwan (3):
  - Site 2352, Kaohsiung City
  - Site 2351, Kaohsiung City
  - Site 2354, Taipei
- Ukraine (14):
  - Site 5264, Chernivtsi
  - Site 5261, Ivano-Frankivsk
  - Site 5258, Ivano-Frankivsk
  - Site 5256, Kharkiv
  - Site 5254, Kharkiv
  - Site 5255, Kherson
  - Site 5263, Kyiv
  - SIte 5252, Kyiv
  - Site 5251, Kyiv
  - Site 5265, Kyiv
  - Site 5259, Poltava
  - Site 5260, Vinnytsia
  - Site 5253, Zaporizhzhya
  - Site 5257, Zaporizhzhya

REFERENCES:
- [Derived] File TM Jr, Alexander E, Goldberg L, Das AF, Sandrock C, Paukner S, Moran GJ. Lefamulin efficacy and safety in a pooled phase 3 clinical trial population with community-acquired bacterial pneumonia and common clinical comorbidities. BMC Pulm Med. 2021 May 8;21(1):154. doi: 10.1186/s12890-021-01472-z. PMID 33964925
- [Derived] Alexander E, Goldberg L, Das AF, Moran GJ, Sandrock C, Gasink LB, Spera P, Sweeney C, Paukner S, Wicha WW, Gelone SP, Schranz J. Oral Lefamulin vs Moxifloxacin for Early Clinical Response Among Adults With Community-Acquired Bacterial Pneumonia: The LEAP 2 Randomized Clinical Trial. JAMA. 2019 Nov 5;322(17):1661-1671. doi: 10.1001/jama.2019.15468. PMID 31560372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to enroll adults with CABP for which oral antibacterial therapy was appropriate. Subjects with PORT score of II, III and IV were eligible. The first subject was randomized in August 2016 and the last subject was randomized in December 2017
Pre-assignment Details: Subjects who met inclusion criteria and did not meet exclusion criteria were randomly assigned to a treatment group. Administration of study drug was expected to occur as soon as possible after the diagnosis of CABP with all Screening/baseline assessments expected to be completed within 24 hours before the first dose of study drug.
Period: Overall Study
Arm/Group | Lefamulin | Moxifloxacin
Started | 370 (Intent to Treat Analysis Set) | 368 (Intent to Treat Analysis Set)
Completed (Completed Study (Late Follow Up Assessment)) | 353 | 354 (Completed Study (Late Follow Up Assessment))
Not Completed | 17 | 14
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 3 | 3
Not completed — Randomized- did not receive study drug | 2 | 0
Not completed — Patient hospitalized | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lefamulin | Moxifloxacin | Total
Number analyzed (Participants) | 370 | 368 | 738
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (16.4) | 57.7 (16.2) | 57.5 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 188 | 351
  Male | 207 | 180 | 387
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 38 | 83
  Not Hispanic or Latino | 325 | 330 | 655
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 17 | 41
  Asian | 49 | 53 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 22 | 41
  White | 274 | 270 | 544
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 6 | 7 | 13
  Romania | 11 | 7 | 18
  Hungary | 13 | 15 | 28
  United States | 11 | 12 | 23
  Philippines | 35 | 36 | 71
  Ukraine | 65 | 63 | 128
  Russia | 31 | 24 | 55
  Spain | 0 | 1 | 1
  South Korea | 12 | 14 | 26
  Latvia | 3 | 0 | 3
  Taiwan | 0 | 1 | 1
  Poland | 4 | 3 | 7
  Mexico | 1 | 3 | 4
  South Africa | 21 | 34 | 55
  Georgia | 22 | 19 | 41
  Bulgaria | 38 | 42 | 80
  Chile | 2 | 2 | 4
  Serbia | 66 | 63 | 129
  Peru | 29 | 22 | 51
Renal Status [Count of Participants; unit: Participants]
  Severe impairment (CrCl <30 mL/min) | 4 | 3 | 7
  Moderate impairment (CrCl 30 to <60 mL/min) | 64 | 70 | 134
  Mild impairment (CrCl 60 to <90 mL/min) | 112 | 117 | 229
  Normal function (CrCl >/= 90 mL/min) | 190 | 178 | 368
Pneumonia Outcomes Research Team (PORT) Risk Class [Count of Participants; unit: Participants] — PORT Risk Class is a clinical prediction rule used to calculate risk of morbidity and mortality among patients presenting with community-acquired pneumonia taking into consideration age, history of comorbid conditions, physical examination findings, and laboratory or radiographic results. PORT Risk Class I is a PORT score of 0-50, II is 51-70, III is 71-90, IV is 91-130 and V is >130 with higher risk class indicating higher risk of morbidity and mortality.
  Participants
    I | 1 | 2 | 3
    II | 183 | 189 | 372
    III | 145 | 133 | 278
    IV | 40 | 42 | 82
    V | 1 | 2 | 3
CURB-65 Score [Count of Participants; unit: Participants] — CURB-65 is a clinical tool used to predict mortality in patients with community acquired pneumonia. The risk of death at 30 days increases as the score increases; a score of 0 indicates the lowest risk of death and a score of 5 indicates the highest risk of death. Defined as confusion of new onset, BUN >19 mg/dL, respiratory rate ≥30 breaths/min, systolic blood pressure <90 mm Hg or diastolic blood pressure ≤60 mm Hg, and age ≥65 years.
  Participants
    0 | 87 | 80 | 167
    1 | 197 | 196 | 393
    2 | 74 | 77 | 151
    3 | 12 | 13 | 25
    4 | 0 | 2 | 2
    5 | 0 | 0 | 0
American Thoracic Society (ATS) Minor Severity Criteria [Count of Participants; unit: Participants] — ATS minor criteria are used to indicate severe community acquired pneumonia and suggests the need for intensive care unit (ICU) level care. Defined as presence of 3 or more of the following 9 criteria at baseline: respiratory rate of 30 breaths/min or greater, oxygen saturation less than 90% or PaO2 less than 60mmHg, blood urea nitrogen level of 20mg/dL or greater, white blood cell count less than 4,000/mm3, confusion, multilobar infiltrates, platelet level less than 100,000 cells/mm3, temperature lower than 36 °C, or systolic blood pressure less than 90mmHg.
  Participants | 31 | 37 | 68
Systemic inflammatory response syndrome (SIRS) Criteria [Count of Participants; unit: Participants] — SIRS is used to define a clinical response to a nonspecific insult of either infectious or noninfectious origin. SIRS is defined as a subject meeting at least 2 or more of the following: Fever of more than 38C (100.4F) or less than 36C (96.8F); heart rate greater than 90 beats/min; respiratory rate greater than 20 breaths/min or PaCO2 less than 32 mm Hg; abnormal white blood cell count (greater than 12,000/microL or less than 4,000/microL or greater than 10% immature band forms)
  Participants | 353 | 342 | 695
Bacteremic [Count of Participants; unit: Participants] | 6 | 9 | 15
Received Single Dose Short-Acting Antibacterial within 72 hrs of Randomization [Count of Participants; unit: Participants] | 77 | 72 | 149

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response (ECR)
Description: ECR was defined as survival with improvement in at least 2 signs and symptoms of CABP (relative to baseline), no worsening of any CABP sign or symptom, and no use of concomitant antibiotics for the treatment of CABP through the ECR assessment
Time Frame: 96 hours +/- 24 hours after first dose of study drug
Population: Intent to Treat Analysis Set: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Lefamulin | Moxifloxacin
Number analyzed (Participants) | 370 | 368
Participants
  Responder | 336 | 334
  Non-responder | 29 | 31
  Indeterminate | 5 | 3
Statistical Analysis 1: Comparison: Lefamulin vs Moxifloxacin; Test type: Non-Inferiority — non-inferiority margin= 10%; Treatment difference = 0.1, 95% CI 2-sided [-4.4 to 4.5] — Difference in percentage of Responders for ECR (Lefamulin - Moxifloxacin). Confidence interval computed using continuity-corrected Z-statistic

2. Secondary Outcome: Investigator's Assessment of Clinical Response (IACR)
Description: IACR was defined as resolution or improvement of a subject's clinical signs and symptoms such that no additional antibacterial therapy was administered for the treatment of the current episode of CABP
Time Frame: IACR was assessed at the Test-of-Cure Visit; 5 to 10 days after last dose of study drug
Population: Modified ITT population: All randomized subjects who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Lefamulin | Moxifloxacin
Number analyzed (Participants) | 368 | 368
Participants
  Success | 322 | 328
  Failure | 44 | 32
  Indeterminate | 2 | 8
Statistical Analysis 1: Comparison: Lefamulin vs Moxifloxacin; Test type: Non-Inferiority — non-inferiority margin = 10%; Treatment difference = -1.6, 95% CI 2-sided [-6.3 to 3.1] — Difference in Percentage of Success for IACR at test of cure visit (Lefamulin - Moxifloxacin). CI computed via Miettinen-Nurminen method, adjusted for prior antibiotic use [Y vs. N] and PORT risk class [III vs. IV/V], using CMH stratum weights
Statistical Analysis 2: Comparison: Lefamulin vs Moxifloxacin; Test type: Non-Inferiority — non-inferiority margain = 10%; Treatment difference = -1.6, 95% CI 2-sided [-6.5 to 3.3] — Difference in percentage of Success for IACR at test of cure visit. Confidence interval computed using a continuity-corrected Z-test

3. Secondary Outcome: Investigator's Assessment of Clinical Response (IACR)
Description: as for outcome 2
Time Frame: IACR was assessed at the Test-of-Cure Visit; 5 to 10 days after last dose of study drug
Population: Clinically Evaluable population: Subset of ITT population having met additional pre-defined criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Lefamulin | Moxifloxacin
Number analyzed (Participants) | 330 | 326
Participants
  Success | 296 | 305
  Failure | 34 | 21
Statistical Analysis 1: Comparison: Lefamulin vs Moxifloxacin; Test type: Non-Inferiority — non-inferiority margain = 10%; Treatment difference = -3.9, 95% CI 2-sided [-8.2 to 0.5] — Difference in percentage of success for IACR at test of cure visit (Lefamulin - Moxifloxacin). CI computed via Miettinen-Nurminen method, adjusted for prior antibiotic use [Y vs. N]; PORT risk class [III vs. IV/V], using CMH stratum weights
Statistical Analysis 2: Comparison: Lefamulin vs Moxifloxacin; Test type: Non-Inferiority — non-inferiority margin = 10%; Treatment difference = -3.9, 95% CI 2-sided [-8.4 to 0.7] — Difference in Percentage of Success for IACR at test of cure visit (Lefamulin - Moxifloxacin). Confidence interval computed using continuity-corrected Z-statistic

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of informed consent through the completion of the Test-of-Cure (TOC) Visit (i.e., 5-10 days after the last dose of study drug). Serious adverse events were recorded from the time of informed consent to the Late Follow-Up Visit (approximately 30 days after the first dose of study drug).
Description: Adverse events are reported for randomized subjects who received at least one dose of study drug (Safety Population). Treatment-emergent adverse events, defined as events occurring after the first dose of study drug, are reported. Adverse events were recorded whether or not they were considered to be study drug related.
Arm/Group | Lefamulin | Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 5/368 | 3/368
Serious Adverse Events (participants affected / at risk) | 17/368 | 18/368
Other Adverse Events (participants affected / at risk) | 61/368 | 12/368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lefamulin (N=368) | Moxifloxacin (N=368)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 2
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Lung Abscess (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 4 | 1
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Tuberculous Pleurisy (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
Nuclear Magnetic Resonance Imaging Brain Abnormal (Investigations) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Embolic Stroke (Nervous system disorders) | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lefamulin (N=368) | Moxifloxacin (N=368)
Diarrhoea (Gastrointestinal disorders) | 45 | 4
Nausea (Gastrointestinal disorders) | 19 | 7
Vomiting (Gastrointestinal disorders) | 12 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data from the study is confidential information. Sponsor has the right to publish first. Thereafter, PI may publish data from the study, but PI must submit the publication to Sponsor for review at least 60 days prior to publication. Sponsor may remove any confidential and/or proprietary information. If Sponsor's publication is not submitted within 12 months after the study, or if Sponsor decides not to publish, PI may publish the data, subject to Sponsor's rights in the agreement.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT02813694/SAP_000.pdf
  • Study Protocol (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT02813694/Prot_001.pdf